CLINICAL TRIAL: NCT03623334
Title: Phase I Study of Accelerated Hypofractionated Image-Guided Radiation Therapy (IGRT) in Patients With Stage II-IV Non-Small Cell Lung Cancer and Poor Performance Status
Brief Title: Phase I Study of Accelerated Hypofractionated Image-Guided Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU 072010-050
Record Dates: First submitted 2018-05-14; First posted 2018-08-09 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Level A: IGRT 3.33Gy x 15 Fractions (Experimental): Image-guided radiation therapy (IGRT) dose of 3.33Gy for 15 fractions (total dose = 50 Gy) which is given over the course of about 3 weeks
  Interventions: Radiation: Image-Guided Radiation Therapy
- Dose Level B: IGRT 3.67Gy x 15 Fractions (Experimental): Image-guided radiation therapy (IGRT) dose of 3.67Gy for 15 fractions (total dose = 55 Gy) which is given over the course of about 3 weeks
  Interventions: Radiation: Image-Guided Radiation Therapy
- Dose Level C: IGRT 4.00Gy x 15 Fractions (Experimental): Image-guided radiation therapy (IGRT) dose of 3.67Gy for 15 fractions (total dose = 60 Gy) which is given over the course of about 3 weeks
  Interventions: Radiation: Image-Guided Radiation Therapy

INTERVENTIONS:
Radiation: Image-Guided Radiation Therapy — Radiotherapy to a potent tumorcidal dose

SUMMARY:
The study is designed to determine whether daily image guidance and motion assessment/control will allow treatment of poor performance status patients with stage II-IV NSCLC, who would benefit from local therapy, with an accelerated course of hypofractionated radiation therapy.

DETAILED DESCRIPTION:
Subjects for this study will be enrolled by the Moncrief Radiation oncology Department at the Simmons Cancer Center.

Primary objective: To escalate the dose of accelerated, hypofractionated, image-guided conformal radiotherapy to a potent tumorcidal dose without exceeding the maximum tolerated dose in treatment of stage ii-iV nSCLC in patients with poor performance status.

Secondary objectives: To evaluate local regional tumor control and overall survival in patients with stage ii-iV nSCLC and poor performance status treated with accelerated, hypofractionated, image-guided conformal radiotherapy.

Schema

number of patients between 7-45 (depending on tolerance)

Patients in each dose cohort will all be treated as a single group for dose escalation. The starting dose will be 3.33 Gy per fraction for 15 fractions (total dose 50 Gy). Subsequent cohorts of patients will receive a higher dose per fraction as follows:

Cohort No. Fractions Dose per fraction (Gy) Total Dose (Gy) No. Patients

1. 15 3.33 50 7-15
2. 15 3.67 55 7-15
3. 15 4.00 60 7-15

Minimum waiting periods will be assigned between each dose cohort to observe toxicity.

Screening Procedures

each study participant will have the following exams, tests or procedure to help determine if they are qualified to be in this study:

Within 8 weeks of enrollment :

* Computed tomographic (CT) with contrast of the lung and upper abdomen. a CT done in conjunction with a Positron emission Tomography (PeT) scan is satisfactory as long as the images are of adequate quality to be interpreted by a radiologist.
* an MRi of the brain with contrast (or CT if MRi is medically contraindicated).
* Complete Blood Count (CBC) with differential
* Charleston Comorbidity index completion

Within 3 days prior to radiotherapy: urine or serum pregnancy test in females of child-bearing capacity.

Within 12 weeks of enrollment:

* Pulmonary function tests including spirometry for forced expiratory volume in 1 second (FeV-1), diffusing capacity (DLCo), and arterial blood gas (Pao-2).

Prior to enrollment on the study: Tissue biopsy or cytology confirming non-small cell lung cancer.

Treatment Protocol treatment must begin within 4 weeks after patient registration to the trial. Patients will receive 15 fractions of radiation. Total dose will depend on the dose cohort of the study (see schema). The starting dose level will be 3.33 Gy per fraction for 15 fractions (total dose [?] 50 Gy).

Patients must not receive other concomitant antineoplastic therapy (including standard fractionated radiotherapy to the chest, chemotherapy, biological therapy, vaccine therapy, and surgery) within a week prior to, during, or within one week after completing hypofractionated image-guided radiation therapy on protocol.

Follow-up Patients will be followed until death.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be willing and capable to provide informed consent to participate in the protocol.
2. Patients must have appropriate staging studies identifying them as AJCC stage II, III or IV non small cell lung cancer, [according to AJCC Staging, 6th edition; see appendix III], or recurrent non small cell lung cancer. Histologic confirmation of cancer will be required by biopsy or cytology.
3. Patients must have the potential for benefit from local therapy (at the discretion of the investigator).
4. Patient must have a Zubrod performance status of 2 or greater Or Patient must have had >10% weight loss in the past 6 months Or Patient is not eligible for concurrent chemoradiation as determined by a Medical Oncologist and Radiation Oncologist
5. Age ≥ 18.
6. The tumor must be ineligible for definitive surgical resection.
7. The tumor must be ineligible for stereotactic body radiation therapy.
8. Patients must have measurable or evaluable disease.
9. Women of childbearing potential and male participants must agree to use an effective method of contraception.
10. Patients must sign study specific informed consent prior to study entry.
11. Patients must complete all required pretreatment evaluations

Exclusion Criteria:

1. Evidence of small cell histology.
2. Tumor eligible for definitive surgical resection.
3. Tumor eligible for definitive stereotactic body radiation therapy.
4. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
5. Chemotherapy given within one week of study registration.
6. Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-10-05 (Actual); Primary Completion 2012-11-02 (Actual); Study Completion 2018-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Timmerman, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level A: IGRT 3.33Gy x 15 Fractions (Total 50 Gy): Image-guided radiation therapy (IGRT) dose which is given over the course of about 3 weeks
  Patients with stage II to IV or recurrent NSCLC and Eastern Cooperative Oncology Group performance status of 2 or greater and not candidates for surgical resection, stereotactic radiation, or concurrent chemoradiation were eligible. Highly conformal radiation therapy was given to treat intrathoracic disease in 15 fractions to a total of 50, 55, or 60 Gy.
- Dose Level B: IGRT 3.67Gy x 15 Fractions (Total 55-Gy ): Image-guided radiation therapy (IGRT) which is given over the course of about 3 weeks
  Patients with stage II to IV or recurrent NSCLC and Eastern Cooperative Oncology Group performance status of 2 or greater and not candidates for surgical resection, stereotactic radiation, or concurrent chemoradiation were eligible. Highly conformal radiation therapy was given to treat intrathoracic disease in 15 fractions to a total of 50, 55, or 60 Gy.
- Dose Level C: IGRT 4Gy x 15 Fractions ( Total 60Gy): 4 Gy per fraction for a total dose of 60 Gy will be tested. Image-guided radiation therapy (IGRT) dose which is given over the course of about 3 weeks
  Patients with stage II to IV or recurrent NSCLC and Eastern Cooperative Oncology Group performance status of 2 or greater and not candidates for surgical resection, stereotactic radiation, or concurrent chemoradiation were eligible. Highly conformal radiation therapy was given to treat intrathoracic disease in 15 fractions to a total of 50, 55, or 60 Gy.
Period: Overall Study
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (Total 50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (Total 55-Gy ) | Dose Level C: IGRT 4Gy x 15 Fractions ( Total 60Gy)
Started | 15 | 21 | 19
Completed | 15 | 21 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level A: IGRT 3.33Gy x 15 Fractions (Total 50Gy): Image-guided radiation therapy (IGRT) does of 3.33Gy for 15 fractions (total dose = 50 Gy) which is given over the course of about 3 weeks
- Dose Level B: IGRT 3.67Gy x 15 Fractions (Total 55Gy): Image-guided radiation therapy (IGRT) dose of 3.67Gy for 15 fractions (total dose = 55 Gy) which is given over the course of about 3 weeks
- Total: Total of all reporting groups
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (Total 50Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (Total 55Gy) | Dose Level C: IGRT 4Gy x 15 Fractions ( Total 60Gy) | Total
Number analyzed (Participants) | 15 | 21 | 19 | 55
Age, Continuous [Median (Full Range); unit: years] | 65 [30 to 84] | 65 [30 to 84] | 65 [30 to 84] | 65 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 11 | 24
  Male | 12 | 11 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity
Description: A dose limiting toxicity (DLT) is defined as treatment-related (definitely and probably, but not possibly related to treatment*) grade 3 adverse events (per CTCAE, v.3.0, with the exception of pulmonary function tests)
Time Frame: 90 days after start of treatment up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy): In this cohort, the starting dose of Image-Guided Radiation Therapy (IGRT) will be 3.33 Gy per fraction for 15 fractions (total dose = 50 Gy).
- Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy): In this cohort, the starting dose of Image-Guided Radiation Therapy (IGRT) will be 3.67 Gy per fraction for 15 fractions (total dose = 55 Gy).
- Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy): In this cohort, the starting dose of Image-Guided Radiation Therapy (IGRT) will be 4.00 Gy per fraction for 15 fractions (total dose = 60 Gy).
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 15 | 21 | 19
Participants | 1 | 1 | 1

2. Secondary Outcome: Number of Participants With Local Regional Tumor Control at 3 Months
Description: Local control is defined as the absence of isolated progression (stable disease or responsive disease at last follow-up) within the primary tumor. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: 3 months
Population: Only convenient sample were included. Those who died, lost to follow-up, refused scans were not included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 9 | 17 | 15
Participants | 4 | 11 | 11

3. Secondary Outcome: Number of Participants With Local Regional Tumor Control at 6 Months
Description: as for outcome 2
Time Frame: 6 months
Population: Only convenient sample were included. Those who died, lost to follow-up, refused scans were not included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 8 | 9 | 10
Participants | 2 | 5 | 8

4. Secondary Outcome: Number of Participants With Local Regional Tumor Control at 9 Months
Description: as for outcome 2
Time Frame: 9 months
Population: Only convenient sample were included. Those who died, lost to follow-up, refused scans were not included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 3 | 5 | 7
Participants | 2 | 4 | 5

5. Secondary Outcome: Number of Participants With Local Regional Tumor Control at 12 Months
Description: as for outcome 2
Time Frame: 12 months
Population: Only convenient sample were included. Those who died, lost to follow-up, refused scans were not included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 1 | 3 | 5
Participants | 1 | 1 | 4

6. Secondary Outcome: Number of Participants With Local Regional Tumor Control at 16 Months
Description: as for outcome 2
Time Frame: 16 months
Population: Only convenient sample were included. Those who died, lost to follow-up, refused scans were not included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 1 | 1 | 3
Participants | 1 | 0 | 2

7. Secondary Outcome: Number of Participants With Local Regional Tumor Control at 20 Months
Description: as for outcome 2
Time Frame: 20 months
Population: Only convenient sample were included. Those who died, lost to follow-up, refused scans were not included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 1 | 1 | 0
Participants | 1 | 0 | 0

8. Secondary Outcome: Overall Survival at 6 Months
Description: Overall survival is defined as participants alive during the research period.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy)
Number analyzed (Participants) | 15 | 21 | 19
Participants | 11 | 13 | 12

ADVERSE EVENTS:
Time Frame: This was collected over a period of 12 months.
Arm/Group | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy
All-Cause Mortality (participants affected / at risk) | 14/15 | 14/21 | 11/19
Serious Adverse Events (participants affected / at risk) | 5/15 | 4/21 | 4/19
Other Adverse Events (participants affected / at risk) | 15/15 | 20/21 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) (N=15) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) (N=21) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy (N=19)
G2 or higher dyspnea (Cardiac disorders) | 5 | 4 | 4
G2 or higher Esophagitis (General disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level A: IGRT 3.33Gy x 15 Fractions (50 Gy) (N=15) | Dose Level B: IGRT 3.67Gy x 15 Fractions (55 Gy) (N=21) | Dose Level C: IGRT 4.00Gy x 15 Fractions (60 Gy (N=19)
≤G2 Esophagitis (General disorders) | 15 | 20 | 18
≤G2 Dyspnea (Cardiac disorders) | 10 | 17 | 15
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Anorexia (Psychiatric disorders) | 3 | 2 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Dysphagia (General disorders) | 3 | 2 | 2
Pain (Nervous system disorders) | 3 | 8 | 12
Anxiety (Nervous system disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Confusion (Nervous system disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Dehydration (Gastrointestinal disorders) | 1 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 7
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypotension (Cardiac disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 4
Neuropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Pneumonia (Infections and infestations) | 4 | 1 | 1 — Pulmonary/ Upper Respiratory Infection: Lung (Pnemonia)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Planned statistical analysis was not able to be performed due to the poor overall survival of the study population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03623334/Prot_SAP_000.pdf